CLINICAL TRIAL: NCT05118932
Title: Examining Effects of Holistic School Enrichment Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00129138
Record Dates: First submitted 2021-10-21; First posted 2021-11-12 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Mindful Movement Intervention (MMI)
Keywords: Mindfulness; Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: All students will be receiving the same single intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindful Movement Intervention (Experimental): The Mindful Movement Intervention (MMI) targets improved attentional, behavioral and emotional regulation through engagement of the motor system and mindful practice in school-age children. For this project, children will participate in the MMI twice a week for 45 minutes a session for the duration of the academic year. The intervention will be held during school hours to make it more accessible to all students and require fewer additional resources.
  Briefly, there are five components that make-up the Mindful Movement Intervention: Biomechanical Warm-ups, Yoga postures, a modified Tai Chi sequence, Imaginative Play, and Reflection.
  One goal of this intervention is to help children to develop the skills needed to cope with naturally occurring changes and to adapt to their environment in a mindful, non-reactive manner. In this context, students are learning to control and manage their attention, behavior and emotion through implicit procedural learning.
  Interventions: Behavioral: Mindful Movement Intervention
- Mindful Movement Intervention Family Based Component (Experimental): In this additional component, participants and their families will have access to monthly Mindful Movement activities intended to reinforce concepts discussed in Mindful Movement class and foster familial relationships. The family-based component will include access to lesson plans and accompanying resources (e.g., videos, worksheets, audio tracks) once a month from October through May, that offer strategies to improve awareness of thoughts, emotions, and body. Families will also be expected to track their adherence to the lesson plans and provide feedback via a survey.
  Interventions: Behavioral: Mindful Movement Intervention
- Mindful Movement Intervention Peer to Peer Mentorship Component (Experimental): In this additional component, participants will have the opportunity to become student instructors and lead younger students in modified instructional classes.
  Interventions: Behavioral: Mindful Movement Intervention
- Mindful Movement Intervention Community Education Component (Experimental): In this additional component, participants will have the option to assist with the development of an instructional video that showcases students in the Mindful Movement program demonstrating mindful movement practices such as breathing techniques, yoga poses, and T'ai Chi movements.
  Interventions: Behavioral: Mindful Movement Intervention

INTERVENTIONS:
Behavioral: Mindful Movement Intervention — There are five components that together make-up the Mindful Movement Intervention: Biomechanical Warm-ups, Yoga postures, modified Tai Chi sequence, Imaginative Play, and Reflection. During the year, participants will learn a "Simplified" Form of a classic Tai Chi sequence. Yoga movements will be used to prepare participants for the nuanced movements of Tai Chi practice, with both Yoga and Tai Chi providing a physical framework in which participants can track their own progress and begin to understand how to better regulate their attention, behavior and emotional responses. Imaginative Play and Reflection Activities are used to stimulate a deeper curiosity in participants about the everyday use and employment of mindfulness practice and to engage participants.

SUMMARY:
The investigators propose to evaluate the efficacy of a Mindful Movement Intervention (MMI) within the Baltimore City Public School (BCPS) system. The goal is to help at-risk youth improve skills important to attentional, behavioral, motor, and emotional control through engagement of mindful movement practices.

To assess the feasibility and efficacy of the program, standardized assessments will be conducted at three time points: the beginning of the school year at the start of the intervention (early September), at the mid-year point (late January), and prior to the end of the school year (early June). During these assessments, participants will be pulled out of their academic classes for brief sessions (1 hour) in which they will complete assessments of attentional, behavioral, motor, and emotional control. At these assessment points, parents and teachers will complete rating forms about the children including assessments of emotional, behavioral, and attention regulation.

Research participants will have the option to reinforce mindful movement practices using a family-based curriculum, participating in peer mentorship, and supporting the development of community educational materials.

ELIGIBILITY:
Inclusion Criteria:

1. Students must be between the ages 7 years, 0 months and 15 years, 11 months, 30 days.
2. Students with a diagnosis of depression, anxiety, autism, oppositional defiant disorder, and post traumatic stress disorder can be included in the research study
3. Students taking stimulant medications and all other psychoactive medications can be included in the research study.
4. Students in general education classrooms with supports, aides, and/or pull-outs

Exclusion Criteria:

1. Diagnosis of...

   * intellectual disability
   * a neurological disorder (e.g., epilepsy, cerebral palsy, traumatic brain injury, Tourette Syndrome)
   * conduct disorder or a recorded history of symptoms consistent with conduct disorder
   * a documented hearing impairment ≥ 25 dB loss in either ear
   * significant learning difficulties that require a special education plan.
2. Students in foster care
3. Students who are or may be pregnant

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Dimensional Assessment of the Evolution of Attention-Deficit/Hyperactivity Symptoms | 9 months
  The Strengths and Weaknesses of ADHD-symptoms and Normal-behavior (SWAN) rating scale has been developed to measure children's attention skills as well as emotional and behavioral regulatory control. The seven-point questionnaire ranges from +3 (far below average) to -3 (far above average).
  Parent and teacher versions of the SWAN will be collected for each participant and subscale and total scores on the SWAN will be assessed at the start of the intervention (month 0), midway through the intervention (month 4) and at the end of the intervention (month 9).
Assessment of the Evolution of Attention-Deficit/Hyperactivity Symptoms | 9 months
  The DuPaul rating scale is used to assess ADHD related behaviors over the past six months. The 18-item scale uses a 4-point Likert scale with 0 = Not at all and 3 = Very Often.
  Parent and teacher versions the DuPaul will be collected for each participant and subscale and total scores on the DuPaul will be assessed at the start of the intervention (month 0), midway through the intervention (month 4) and at the end of the intervention (month 9).

SECONDARY OUTCOMES:
Evolution of Executive Functioning Skills | 9 months
  The evolution of executive functioning skills will be assessed with the Delis-Kaplan Executive Function System (DKEFS) Trails.
  The DKEFS number-letter switching score will be assessed at the start of the intervention (month 0), midway through the intervention (month 4) and at the end of the intervention (month 9).
Evolution of Inhibitory Control | 9 months
  The evolution of inhibitory control will be assessed with a Simple Go/No-Go task.
  The commission error rate and reaction time variability on the Go/No-Go task will be assessed at the start of the intervention (month 0), midway through the intervention (month 4) and at the end of the intervention (month 9).

OTHER OUTCOMES:
Evolution of Motor Function | 9 months
  The evolution of motor function will be assessed by the Physical and Neurological Examination for Subtle Signs (PANESS). The 32 item motor exam includes possible scores ranging from 0 to 105, with higher scores indicating worse motor function.
  The total score, overflow movement score, and dysrhythmia score from the PANESS will be assessed at the start of the intervention (month 0), midway through the intervention (month 4) and at the end of the intervention (month 9).
Evolution of Motor Persistence | 9 months
  The evolution of motor persistence will be assessed by the Developmental Neuropsychological Assessment (NEPSY) Statue. During a 75-second time period, children will attempt to ignore sound distractors while maintaining a body position. The total score ranges from 0 to 30 with higher scores indicating better performance.
  The total score from the NEPSY statue will be assessed at the start of the intervention (month 0), midway through the intervention (month 4) and at the end of the intervention (month 9).
Evolution of Motor Control | 9 months
  The evolution of motor control will be assessed by the Lateral Gaze Fixation. Students will be timed until 30 seconds with longer times indicating better performance.
  The total time from the Lateral gaze fixation will be assessed at the start of the intervention (month 0), midway through the intervention (month 4) and at the end of the intervention (month 9).
Evolution of Response Inhibition | 9 months
  The evolution of response inhibition will be assessed with administration of the flanker task.
  Incongruent error rate and reaction time variability from the flanker task will be assessed at the start of the intervention (month 0), midway through the intervention (month 4) and at the end of the intervention (month 9).
Evolution of Child-Reported Emotion Regulation | 9 months
  The evolution of child-reported emotion regulation will be assessed by the Social Emotional Assets and Resilience Scales Child-Report (SEARS-C) short form questionnaire. This questionnaire is a 12-item scale that uses a 4-point Likert scale with 0= Never and 3-Always.
  The subscale and total score on the SEARS-C questionnaire will be assessed at the start of the intervention (month 0), midway through the intervention (month 4) and at the end of the intervention (month 9).
Evolution of Caregiver-Reported Emotion Regulation | 9 months
  The evolution of caregiver-reported emotion regulation will be assessed by the Social Emotional Assets and Resilience Scales (SEARS). This questionnaire is a 35-item scale that uses a 4-point Likert scale with 0= Never and 3-Always.
  The subscale and total score on the SEARS questionnaire will be assessed at the start of the intervention (month 0), midway through the intervention (month 4) and at the end of the intervention (month 9).
Assessment of Caregiver-Family Quality of Life | 9 months
  The assessment of family quality of life will be measured by the Family Quality of Life Scale (FQOL Scale). This questionnaire is a 25-item scale that uses a 5-point Likert scale with 1= Very dissatisfied, 3= Neither satisfied nor dissatisfied, and 5= Very satisfied.
  The subscale and total score on the FQOL questionnaire will be assessed at the start of the intervention (month 0) and at the end of the intervention (month 9).
Evolution of Child-Reported Impulsivity and Risk-Taking Behavior | 9 months
  The evolution of child-reported impulsivity and risk-taking behavior will be assessed by the UPPS (urgency, premeditation, perseverance, and sensation seeking) Impulsivity Scale, child version. This questionnaire is a 40-item scale that uses a 4-point Likert scale with 1=strongly disagree to 4=strongly agree.
  The subscale and total score on the UPPS questionnaire will be assessed at the start of the intervention (month 0), midway through the intervention (month 4), and at the end of the intervention (month 9).
Evolution of Child-Reported Tolerance to Uncertainty | 9 months
  The evolution of child-reported tolerance to uncertainty will be assessed by the intolerance of uncertainty scale for children (IUSC). This questionnaire is a 27-item scale that uses a 5-point Likert scale with 1=not at all, 3= somewhat, 5= very much.
  The subscale and total score on the IUSC questionnaire will be assessed at the start of the intervention (month 0), midway through the intervention (month 4), and at the end of the intervention (month 9).

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Mostofsky, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (2):
- United States (2):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - City Neighbors Charter School, Baltimore, Maryland